CLINICAL TRIAL: NCT03829969
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Compare Toripalimab Injection (JS001) Combined With Standard Chemotherapy Versus Placebo Combined With Standard Chemotherapy in Treatment of Advanced or Metastatic Esophageal Squamous Cell Cancer (ESCC) Without Previous Systemic Chemotherapy
Brief Title: Toripalimab or Placebo With Paclitaxel and Cisplatin in Esophageal Squamous Cell Carcinoma
Acronym: JUPITER06
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-021-III-ESCC
Record Dates: First submitted 2019-01-17; First posted 2019-02-04 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-02

CONDITIONS: Advanced or Metastatic Esophageal Squamous Cell Cancer Without Previous Systemic Chemotherapy
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Toripalimab (Experimental): Toripalimab combine with paclitaxel and cisplatin
  Interventions: Biological: Toripalimab
- placebo (Placebo Comparator): Placebo combine with paclitaxel and cisplatin
  Interventions: Biological: Toripalimab

INTERVENTIONS:
Biological: Toripalimab — TORIPALIMAB INJECTION(JS001 ) combine with chemotherapy or placebo combine with chemotherapy
  Other Names: JS001, TAB001

SUMMARY:
This is one randomized, double-blind, multi-center, placebo-controlled phase III study. The objective of this study is to compare the effectiveness and safety of JS001 combined with paclitaxel and cisplatin(TP regimen )with placebo combined with TP regimen in patients with advanced or metastatic Esophageal Squamous Cell Carcinoma(ESCC )who have not received systemic chemotherapy previously.

ELIGIBILITY:
Inclusion Criteria： Inclusion criteria for oesophageal cancer Histologically or cytologically diagnosed locally advanced / recurrent or metastatic ESCC without radical treatment; No prior systemic anti-tumor therapy for recurrent or metastatic tumor. No recurrence at least 6 months from the end of last treatment in the patients previously receiving adjuvant, neoadjuvant chemotherapy/radiotherapy/chemoradiotherapy and radical therapy for non-metastatic disease (No recurrence at least 12 months from the end of last treatment in the patients previously receiving adjuvant chemotherapy/chemoradiotherapy with TP regimen); No risk of major hemorrhage or esophageal fistula, for example, large ulcer at the lesion is considered as the risk for major hemorrhage and esophageal fistula, the patient is not suitable to be enrolled. Subjects with tumor directly invading adjacent organs such as the aorta or trachea (T4b disease) should be closely assessed for risk of hemorrhage or fistula and consult the sponsor prior to enrollment.

General requirements for inclusion:

Signed informed consent; Male or female aged 18 to 70 years ECOG score 0 or 1; Expected survival longer than 3 months; Agreement upon providing previously reserved tumor tissue specimen or biopsied tumor lesion tissue for biomarker analysis.

At least one measurable lesion in accordance with RECIST 1.1 (only when clear progression of disease occurs after radiotherapy for the previously irradiated lesion, the lesion can be used as measurable lesion).

Good organ function level:

Hematology: neutrophil ≥1.5×10^9/L, hemoglobin ≥9 g/dL and platelet ≥100×10^9/L.

Hepatic function: bilirubin ≤1.5 time of upper limit of normal (ULN) (patients who are known to have Gilbert disease and serum bilirubin level ≤3 times of ULN can be enrolled), AST and ALT ≤2.5 times of ULN (in case of hepatic metastasis, AST /ALT≤5 times of ULN), and alkaline phosphatase≤3 times of ULN (in case of hepatic or bone metastasis, ALP≤5 times of ULN); albumin ≥3g / dL; International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5 x ULN.

Renal function: serum creatinine ≤1.5 × ULN or estimated glomerular filtration rate in accordance with Cockcroft-Gault formula: creatinine clearance ≥60 mL/min ((140 - age)x(weight，kg)x(0.85，for women))/(72 x(serum creatinine，mg/dL))

Or:

((140 - age)x(weight，kg)x(0.85，for women))/(0.818 x(serum creatinine，μmol/L))

Women who meet the following criteria are eligible to be included and participate in the study:

No childbearing potential (e.g., physiologically infertile), women meeting any one of the following conditions:

Having undergone uterectomy, Having undergone bilateral oophorectomy (oophorectomy), Having undergone ligation of bilateral fallopian tubes, or Postmenopause (total duration of menopause ≥1 year).

Having childbearing potential, serum pregnancy test negative at screening (within 7 days prior to the first dose of study drug), and adequate contraceptive measures taken prior to entry in the study and throughout the study, until 60 days after the last dose of the study drug. The adequate contraceptive measure taken continuously in accordance with the instruction on the contraceptive product and physician's guidance is defined as below:

Any intrauterine device confirmed to have a failure rate for contraception less than 1% per year Dual barrier contraception is defined as the condom with spermicidal gel, foam, suppository or film; or diaphragma with spermicide; or male condom and diaphragma.

Exclusion Criteria

Cancer-specific exclusion criteria:

Active or untreated CNS metastasis determined through CT or magnetic resonance imaging (MRI) evaluation in screening period and previous radiological evaluation (e.g., brain or leptomeningeal metastasis). Patients who have received previous treatment of brain or meningeal metastases, who have been stabilized for at least 2 months and discontinued systemic hormone therapy (> 10 mg/d of prednisone or equivalent) for > 4 weeks prior to randomization; Uncontrolled tumor related pain; Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage (once per month or more frequent); indewlling catheter (e.g. PleurX®) is allowed; Uncontrollable or symptomatic hypercalcemia (ionized calcium>1.5 mmol/L or calcium >12 mg/dL or corrected serum calcium >ULN); History of malignant tumors except esophageal cancer within 5 years prior to randomization, but except the malignant tumors that risk of metastasis or death can be neglected [e.g., expected 5-year survival rate> 90%], and are expected to be cured after treatment, for example, appropriately treated carcinoma in situ of cervix, basal or squamous cell skin cancer, local prostate cancer treated with radical operation, and ductal carcinoma in situ treated with radical operation; Palliative Radiotherapy within 4 weeks prior to enrollment, or radiopharmaceutical therapy within 8 weeks, however, except locally palliative radiotherapy for bone metastatic lesions; in case of symptomatic lesion suitable for palliative chemotherapy, the therapy should be given prior to enrollment. The effect of previous radiotherapy has been recovered. The shortest recovery period is not required; Subjects with bone metastases of multiple vertebra are prone to fractures and may cause risk of paraplegia, except for Subjects who are assessed as stable and do not need to be treated for the time being evaluated by a specialist.

Subjects with advanced tumors spreading to vital organs and being in risk of developing life-threatening complications in the short term ( eg. metastatic disease burden of liver ≥ 50% of total liver volume).

Subjects with known complete obstruction under endoscopy requiring interventions or surgery to remove obstruction and who have undergone tracheal or esophageal stenting; Subjects whose BMI are less than 17.5, or body weight decrease >10% within 2 months prior to first dose of study treatment (considering changes of massive pleural effusion and ascites) or with severe malnutrition as indicated by other indicators.

General medical exclusion criteria:

Women who are pregnant or lactating, or plan to be pregnant during the study; History of serious allergic reaction, anaphylactoid or other hypersensitive reactions to chimeric or humanized antibody or fusion protein; Known allergy or hypersensitivity to the biological products manufactured from Chinese hamster ovary cells or any component of JS001 preparation; History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-related vascular thrombosis, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, glomerulonephritis; Patients with hypothyroidism who receive stable-dose thyroid hormone replacement therapy can be enrolled in this study (the replacement therapy for hypothyroidism is seen in Appendix 6); Patients with type I diabetes whose blood glucose can be controlled through stable-dose insulin can be enrolled in this study;

Patients with eczema, psoriasis, chronic lichen simplex or only the dermatological manifestations of vitiligo (e.g., patients with psoriatic arthritis will be excluded from the study) are allowed to be enrolled in this study if they meet the following conditions:

The coverage area of rashes must be lower than 10% of body surface area (BSA); The disease has been sufficiently controlled at baseline and only low-potency topical steroid therapy is needed; No acute exacerbation of underlying diseases in the past 12 months [no need of PUVA (Psoralen plus ultraviolet A radiation), methotrexate, retinol, biological preparation, oral calcineurin inhibitor, high-potency or oral steroid therapy].

History of idiopathic pulmonary fibrosis, organized pneumonia (e.g., obliterative bronchiolitis), drug induced pneumonia, idiopathic pneumonia interstitial pneumonia or evidence of active pneumonia found during chest CT scanning for screening; Patients with positive result of human immunodeficiency virus (HIV) test

Patients with hepatitis B (known positive HBV surface antigen HBsAg and HBV DNA ≥1000 cps/ml or 200 IU/ml or higher than upper limit of normal at each study site) or hepatitis C:

Subjects with previous hepatitis B virus (HBV) infection can be included in this study. Such subjects must undergo HBV deoxyribonucleic acid (DNA) testing prior to randomization, and can participate in this study only when HBV DNA is negative (HBV DNA ˂1000 cps/mL or 200 IU/mL or below the upper limit of its normal value); In patients with positive hepatitis C virus (HCV) antibody, only the patients with negative polymerase chain reaction (PCR) HCV ribonucleic acid (RNA) can participate in this study.

Patients with active pulmonary tuberculosis (clinical diagnosis includes clinical history, physical examination and radiological findings, as well as the TB test performed in accordance with local medical routines); Serious infection within 4 weeks prior to randomization, including but not limited to the infection complications, bacteremia and severe pneumonia requiring hospitalization; Oral or intravenous antibiotics within two weeks prior to randomization; patients receiving preventive antibiotic therapy (e.g., for prevention of urinary tract infection or prevention of exacerbation of chronic obstructive pulmonary disease) can be enrolled.

Important cardiovascular diseases, e.g., heart disease defined by New York Heart Association (Grade II or above), myocardial infarction within three months prior to randomization, unstable arrhythmia, unstable angina pectoris, cerebrovascular accident or transient cerebral ischemic attack; patients with known coronary artery disease, congestive heart failure not meeting the above criteria or left ventricular ejection fraction < 50% must receive the regimen that is considered by the attending physician as the optimal for stabilizing therapy, and can consult a cardiologist when necessary; Major surgery (except for diagnostic operation) within 28 weeks prior to randomization or expected major surgery during the study; Previous allogeneic bone marrow transplantation or solid organ transplantation. Use of attenuated live vaccine within 4 weeks prior to randomization, or plan to use such attenuated live vaccine during the study Any other disease, metabolic disorder, physical examination finding or abnormal laboratory examination, with the reason to suspect that it can lead to contraindicated use of the investigational product, or affect reliability of the study results, or place the patient at high risk;

Exclusion criteria related to medications:

Patients who have previously received any approved Chinese patent medicine as anti-tumor indication within 2 weeks before first dose of study drug; Subjects treated with other investigational product or participation in the clinical study for other therapeutic objectives within 28 days prior to randomization (including signature of ICF for other trials, and failure of screening); Previous use of immune checkpoint blocking therapy, for example, anti-programmed death receptor -1 (anti-PD-1) and anti-PD-L1 antibody and other therapeutic antibody; Use of systemic immunostimulator therapy [including but not limited to interferon (IFN) or interleukin-2] within 2 weeks or 5 half-lives (t1/2) prior to randomization, whichever comes later; vaccination of cancer vaccine is allowed in previous treatment; Use of systemic immunosuppressive drugs (>10 mg/d Prednisone or equivalent drug) within two weeks prior to randomization, including but not limited to Prednisone, Cyclophosphamide, azathioprine, methotrexate, thalidomide and tumor necrosis factor (TNF); Patients who have received short-term, low-dose, systemic immunosuppressant (e.g., one single dose of Dexamethasone for nausea) can participate in this study after discussion by investigators and medical monitor and approval by medical monitor; Patients who use inhaled corticosteroids for treatment of chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for treatment of orthostatic hypotension and low-dose glucocorticoid (≤10mg /d Prednisone or equivalent drug) supplement for treatment of hypoadrenocorticism can be enrolled.

Patients who have previously received the hematopoietic growth factors (e.g. granulocyte colony-stimulating factor (G-CSF) and erythropoietin) or blood transfusion within 2 week before randomization.

Exclusion criteria related to chemotherapy:

History of allergy to cisplatin, carboplatin or other platinum-based compounds; Grade 2 or above peripheral neuropathy in accordance with common terminology criteria for adverse event (CTCAE) v5.0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Prof, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Toripalimab | Placebo
Started | 257 | 257
Completed | 257 | 257
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Toripalimab | Placebo | Total
Number analyzed (Participants) | 257 | 257 | 514
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 156 | 163 | 319
  >=65 years | 101 | 94 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.30 (8.04) | 60.90 (7.30) | 61.1 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 77
  Male | 217 | 220 | 437
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 257 | 257 | 514
Region of Enrollment [Number; unit: participants]
  China | 257 | 257 | 514

OUTCOME MEASURES:

1. Primary Outcome: PFS((Progression-Free Surviv)
Description: To evaluate the differences in PFS following JS001 in combination with TP regimen compared to placebo in combination with TP regimen in all randomized patient population with advanced or metastatic ESCC who had not previously received systemic chemotherapy (as assessed by blinded independent central review [BICR] per RECIST 1.1 criteria).
Time Frame: PFS: up to 2years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 132 | 164
months | 5.7 [5.6 to 7.0] | 5.5 [5.2 to 5.6]

2. Primary Outcome: OS (Overall Survival)
Description: To evaluate the differences in OS following JS001 in combination with TP regimen compared to placebo in combination with TP regimen in all randomized patient population with advanced or metastatic ESCC who had not previously received systemic chemotherapy (as assessed by blinded independent central review [BICR] per RECIST 1.1 criteria)
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 172 | 195
months | 17.7 [14.6 to 20.8] | 12.9 [11.6 to 14.1]

3. Secondary Outcome: ORR(Overall Response Rate:BICR)
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy, as measured by blind independent review committee BIRC and investigator-assessed overall response rate (ORR), daccording to RECIST v1.1; ORR:Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 2 approximately years
Measure: Count of Participants; unit: Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 257 | 257
Participants | 178 | 134

4. Secondary Outcome: DCR(Disease Control Rate:BICR )
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy, as measured by blind independent review committee BIRC and investigator-assessed disease control rate (DCR) according to RECIST v1.1 DCR is defined as the proportion of patients with the best efficacy of CR or PR or SD.
Time Frame: Up to 2 approximately years
Measure: Count of Participants; unit: Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 257 | 257
Participants | 229 | 211

5. Secondary Outcome: DOR(Duration of Response: Recist 1.1,BICR )
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy, as measured by blind independent review committee BIRC and investigator-assessed duration of response (DoR) according to RECIST v1.1 DOR is defined as the time from first documented response to first documented evidence of disease progression or to death, whichever comes first.
Time Frame: Up to 2 approximately years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 178 | 134
months | 5.6 [4.4 to 8.7] | 4.2 [4.2 to 4.4]

6. Secondary Outcome: TTR(Time to Initial Response:BICR )
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy, as measured by blind independent review committee BIRC and investigator-assessed Time to initial Response (TTR) according to RECIST v1.1 TTR is defined as the time from randomization to the first recorded response (CR or PR).
Time Frame: Up to 2 approximately years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 178 | 134
months | 1.4 [1.4 to 1.5] | 1.4 [1.4 to 1.4]

7. Secondary Outcome: PFS
Description: To evaluate the efficacy of JS001 plus chemotherapy compared with placebo plus chemotherapy，as measured by investigator-assessed progression free survival (PFS) according to RECIST v1.1
Time Frame: Up to 2 approximately years
Measure: Count of Participants; unit: Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 257 | 257
Participants | 128 | 167

8. Secondary Outcome: PFS Rate:BICR
Description: 1 years PFS rate
Time Frame: Up to 1 years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 132 | 164
Percentage of Participants | 27.8 [20.4 to 35.8] | 6.1 [2.2 to 12.6]

9. Secondary Outcome: OS Rate
Description: 2 years OS rate
Time Frame: up to 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 172 | 195
Percentage of Participants | 39.1 [33.1 to 45.0] | 27.1 [21.7 to 32.7]

10. Secondary Outcome: PFS Assessed Per irRECIST
Description: To evaluate PFS of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST
Time Frame: From date of randomization, until disease progression , loss of clinical benefit ,withdrawal of consent, death, or study termination by the Sponsor, whichever occurs first. Up to 2 approximately years
Measure: Count of Participants; unit: Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 257 | 257
Participants | 128 | 160

11. Secondary Outcome: ORR Assessed Per irRECIST
Description: To evaluate ORR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 257 | 257
Participants | 180 | 136

12. Secondary Outcome: DoR Assessed Per irRECIST:BICR
Description: To evaluate DOR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST
Time Frame: From date of response until progressive disease. Up to 2 approximately years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 180 | 136
months | 5.6 [4.4 to 8.7] | 4.2 [4.2 to 4.4]

13. Secondary Outcome: DCR Assessed Per irRECIST
Description: To evaluate DCR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST
Time Frame: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 257 | 257
Participants | 232 | 218

14. Secondary Outcome: TTR Assessed Per irRECIST:BICR
Description: To evaluate TTR of JS001 plus chemotherapy compared with placebo plus chemotherapy according to irRECIST
Time Frame: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Toripalimab | Placebo
Number analyzed (Participants) | 180 | 136
months | 1.4 [1.4 to 1.5] | 1.4 [1.4 to 1.4]

15. Secondary Outcome: Patient-Reported Outcomes Collected Via the EORTC QLQ-C30
Description: To evaluate the quality of life (QoL) following JS001 in combination with TP regimen compared to placebo in combination with TP regimen in all randomized population.
Time Frame: as for outcome 10
Reporting Status: Not Posted

16. Secondary Outcome: Patient-Reported Outcomes Collected Via the EORTC QLQ-OES18
Description: as for outcome 15
Time Frame: as for outcome 10
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to approximately 49 months
Description: Safety data are based on the 23 February 2023 cut-off date
Arm/Group | Toripalimab | Placebo
All-Cause Mortality (participants affected / at risk) | 174/257 | 198/257
Serious Adverse Events (participants affected / at risk) | 93/257 | 74/257
Other Adverse Events (participants affected / at risk) | 255/257 | 255/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Toripalimab (N=257) | Placebo (N=257)
Gastrointestinal disorder (Gastrointestinal disorders) | 26 | 25
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 19 | 14
Infectious and infectious (Infections and infestations) | 20 | 9
General disorders (General disorders) | 17 | 13
Respiratory ,thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 | 10
Hetapobiliary disorders (Hepatobiliary disorders) | 8 | 5
Injury，poisoning and procedural complications (Injury, poisoning and procedural complications) | 4 | 2
Sikn and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 | 1
Cardica disorders (Cardiac disorders) | 5 | 1
Investigations (Investigations) | 3 | 1
Renal and urinary disorders (Renal and urinary disorders) | 4 | 1
Vascular disorders (Vascular disorders) | 3 | 2
Nervous system disorders (Nervous system disorders) | 3 | 5
Endorcrine disorders (Endocrine disorders) | 4 | 0
Immune system disorders (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Toripalimab (N=257) | Placebo (N=257)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 234 | 228
gastrointestinal disors (Gastrointestinal disorders) | 201 | 202
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 189 | 194
Investigations (Investigations) | 166 | 152
General disorders (General disorders) | 166 | 152
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 137 | 121
Nervous system disorders (Nervous system disorders) | 118 | 122
Respiratory，thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 104 | 82
Musculoskeletal and connective disorders (Musculoskeletal and connective tissue disorders) | 81 | 77
Infections and infestations (Infections and infestations) | 69 | 53
Renal and urinary disorders (Renal and urinary disorders) | 50 | 52
Cardiac disorders (Cardiac disorders) | 41 | 21
Psychiatric disorders (Psychiatric disorders) | 35 | 30
Vascular disorders (Vascular disorders) | 33 | 35
Endocrine disorders (Endocrine disorders) | 43 | 22
Hepatobiliary disorders (Hepatobiliary disorders) | 20 | 15
Injury，poisoning and procedural complications (Injury, poisoning and procedural complications) | 10 | 6
Ear and labyrinth disorders (Ear and labyrinth disorders) | 8 | 6
Immune system disorders (Immune system disorders) | 9 | 8
Reproductive system and breast disorders (Reproductive system and breast disorders) | 6 | 2
Eye disorders (Eye disorders) | 5 | 3
Neoplasms benign，malignant and unspecified（incl cysts and polys） (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT03829969/Prot_SAP_000.pdf